CLINICAL TRIAL: NCT07109336
Title: Development and Prospective Validation of a Heterogeneous Treatment Effect-Based Decision Model for Transarterial Chemoembolization Combined With or Without Atezolizumab Plus Bevacizumab in Unresectable Hepatocellular Carcinoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Jian Lu, Prof., Zhongda Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISMIO2501
Record Dates: First submitted 2025-07-22; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: HCC - Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heterogeneous Treatment Effect-Based Decision Model (Active Comparator): Participations receiving TACE alone or TACE combined with Atezolizumab plus Bevacizumab decsided by Heterogeneous Treatment Effect-Based Decision Model
  Interventions: Device: Heterogeneous Treatment Effect-Based Decision Model
- TACE combined with Atezolizumab plus Bevacizumab (Active Comparator): Participations all receiving TACE combined with Atezolizumab plus Bevacizumab
  Interventions: Device: Heterogeneous Treatment Effect-Based Decision Model

INTERVENTIONS:
Device: Heterogeneous Treatment Effect-Based Decision Model — Heterogeneous Treatment Effect-Based Decision Model

SUMMARY:
Unresectable hepatocellular carcinoma (uHCC) constitutes a significant health burden in the Asia-Pacific (APAC) region, particularly in China, where it is frequently associated with hepatitis B virus (HBV) infection and diagnosed at advanced stages.

Transarterial chemoembolization (TACE) remains the standard treatment for intermediate-stage hepatocellular carcinoma (HCC), though its effectiveness diminishes in unresectable HCC (uHCC) with intermediate-to-high tumor burden. The IMbrave150 trial established atezolizumab plus bevacizumab (Atezo+Bev) as a superior alternative to sorafenib, demonstrating significant survival advantages in uHCC. Given the marked heterogeneity of intermediate-stage HCC, TACE may not benefit all patients equally. The TALENTACE study investigated on-demand TACE combined with Atezo+Bev versus TACE alone in treatment-naïve uHCC patients with intermediate-to-high tumor burden across China and Japan. Results revealed a statistically significant and clinically meaningful improvement in the primary endpoint, TACE- progression-free survival (PFS), though overall survival (OS) remained immature at the time of analysis.

This situation establishes a critical and unmet need for randomized controlled trials (RCTs) combined with extensive real-world evidence (RWE) to facilitate the assessment of individualized treatment heterogeneity and provide precise treatment recommendations in China and select Asia-Pacific regions.

ELIGIBILITY:
Inclusion Criteria:

* • Aged≥18 years

  * Initiated first-line Atezo+Bev.
  * Eligible for TACE treatment or received at least one TACE within ±2 months of Atezo+Bev initiation (before Atezo+Bev start, anytime during Atezo+Bev therapy, or after Atezo+Bev discontinuation).
  * Clinically or pathologically diagnosed uHCC before or at the initiation of Atezo/Bev.The evidence of being diagnosed as "unresectable" may include but is not limited to below:

"Unresectable" or "advanced" directly documented in the medical records History of extrahepatic metastasis as evidenced clinically or by radiology, histology or cytology OR China Liver Cancer (CNLC) Stage IIIb

* At least one visit record after the initiation of Atezo+Bev
* No prior systemic therapy for HCC, especially immunotherapy
* No prior locoregional therapy to the target lesion(s)
* At least one measurable untreated lesion
* ECOG Performance Status of 0-2

Exclusion Criteria:

* • Evidence of extrahepatic spread (EHS)

  * Participating in interventional clinical trials.
  * Being a candidate for curative treatments
  * Any condition representing a contraindication to TACE as determined by the investigators
  * Active or history of autoimmune disease or immune deficiency
  * Untreated or incompletely treated esophageal and/or gastric varices with bleeding or high risk for bleeding
  * A prior bleeding event due to esophageal and/or gastric varices within 6 months prior to initiation of study treatment
  * Evidence of bleeding diathesis or significant coagulopathy
  * Missing critical baseline or outcome data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 790 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | From date of randomization until the date of death from any cause, whichever came first, assessed up to 24 months
  defined as time from index date to death from any cause.

SECONDARY OUTCOMES:
TACE-PFS | From index date to untreatable progression or TACE failure/refractoriness or any cause of death, whichever occurs first, assessed up to 10 months
  defined as the time from index date to untreatable progression or TACE failure/refractoriness or any cause of death, whichever occurs first.
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 10 months
  defined as the time from index date to the first occurrence of disease progression or death from any cause (whichever occurs first), as determined by the investigator according to RECIST v1.1 or mRECIST.
DoR | From the first occurrence of a documented objective response to disease progression or death from any cause (whichever occurs first), assessed up to 10 months
  defined as the time from the first occurrence of a documented objective response to disease progression or death from any cause (whichever occurs first).
TTP | From index date to unTACE able progression or TACE failure/refractoriness (as defined above), assessed up to 10 months
  defined as the time from index date to unTACE able progression or TACE failure/refractoriness (as defined above).
EHS | From index date to the first evidence of Extrahepatic Spread, assessed up to 10 months
  defined as the time from index date to the first evidence of Extrahepatic Spread.